CLINICAL TRIAL: NCT02116387
Title: Traditional Rehabilitation Versus Rehabilitation With the Imoove® Device for Spinal Musculoskeletal Disorders: a Randomised Controlled Trial
Brief Title: Traditional Rehabilitation Versus Rehabilitation With the Imoove® Device for Spinal Musculoskeletal Disorders
Acronym: IMOOVE IT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AOI/2012/AD-01; 2013-A00743-42 (Other: RCB number)
Record Dates: First submitted 2014-04-15; First posted 2014-04-16 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-01

CONDITIONS: Lower Back Pain
Keywords: Proprioception
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Routine Physical Therapy (Active Comparator): Patients randomized to this arm will follow a classic, routine, physical therapy program.
  Intervention: Routine Physical Therapy
  Interventions: Other: Routine Physical Therapy
- I-Moove Physical Therapy (Experimental): Patients randomized to this arm will follow a physical therapy program using the I-Moove device.
  Intervention: I-Moove Physical Therapy
  Interventions: Device: I-Moove Physical Therapy

INTERVENTIONS:
Other: Routine Physical Therapy — Patients randomized to this arm will participate in a classic physical therapy program (15 weeks, a total of 15 sessions).
  Arms: Routine Physical Therapy
Device: I-Moove Physical Therapy — Patients randomized to this arm will participate in a physical therapy program using the I-Moove device (15 weeks, a total of 15 sessions).
  Arms: I-Moove Physical Therapy

SUMMARY:
The main objective of this study is to evaluate in patients with chronic low back pain (lasting for more than 3 months and not postoperative) the effect of an instrumental rehabilitation using the I-Moove ® device compared to a conventional physiotherapy rehabilitation for ambulatory postural stability (mean and standard deviation of excursions from the center of gravity) without visual control, 6 weeks after the start of the rehabilitation protocol. We focus on the relative variation between the values obtained on day 0 versus 6 weeks, via measures performed on a force platform. The results will be stratified into 3 age groups (18-39 years, 40-60 years and over 60 years).

DETAILED DESCRIPTION:
The secondary objectives of this study are to evaluate and compare the two physical therapy techniques at 6 weeks and 6 months after the start of the rehabilitation protocol in terms of:

A - improving postural stability and visual control on an unstable surface (with and without visual control)

B - improving levels of abdominal strength (Ito test) and erector spinae (Sørensen test)

C - the impact of back pain on daily life using questionnaires (Dallas, Québec, FABQ and Tampa questionnaires/scores)

D - Improvement of pain (Visual Analog Scale),

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient is available for 6 months of follow-up
* Patients with pain in the lumbar spine (low back pain) for at least 3 months, not in connection with an operation

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient will have difficulties with follow-up (the patient is about to move, or isn't motivated)
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient is pregnant, parturient, or breastfeeding
* The patient has already participated in a dynamic physical therapy program
* The patient has a contraindication for a treatment used in this study
* The patient has had surgery in the past year
* The patient has a pathology that can interfere with the physical therapy regimen (heart failure, respiratory failure, major orthopedic problems)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-07-04 (Actual); Primary Completion 2018-06-28 (Actual); Study Completion 2018-06-28 (Actual)

PRIMARY OUTCOMES:
Change in postural stability on the platform, eyes closed | Baseline to 6 weeks

SECONDARY OUTCOMES:
Change in postural stability on the platform, eyes closed | Baseline to 6 months
Change in postural stability on the platform, eyes open | Baseline to 6 weeks
Change in postural stability on the platform, eyes open | Baseline to 6 months
Change in postural stability on the platform, eyes open and with an unstable surface | Baseline to 6 weeks
Change in postural stability on the platform, eyes open and with an unstable surface | Baseline to 6 months
Change in postural stability on the platform, eyes closed and with an unstable surface | Baseline to 6 weeks
Change in postural stability on the platform, eyes closed and with an unstable surface | Baseline to 6 months
Abdominal endurance: Ito test | Baseline (day 0)
Abdominal endurance: Ito test | 6 weeks
Abdominal endurance: Ito test | 6 months
Sorensen test | Baseline (day 0)
Sorensen test | 6 weeks
Sorensen test | 6 months
Dallas questionnaire | Baseline (day 0)
Dallas questionnaire | 6 weeks
Dallas questionnaire | 6 months
Quebec questionnaire | Baseline (day 0)
Quebec questionnaire | 6 weeks
Quebec questionnaire | 6 months
FABQ questionnaire | Baseline (day 0)
FABQ questionnaire | 6 weeks
FABQ questionnaire | 6 months
Tampa Score | Baseline (day 0)
Tampa Score | 6 weeks
Tampa Score | 6 months
Visual analog scale for pain | Baseline (day 0)
  ranging from 0 to 10
Visual analog scale for pain | 6 weeks
  ranging from 0 to 10
Visual analog scale for pain | 6 months
  ranging from 0 to 10

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Dupeyron, MD, PhD, Study Director — Centre Hospitalier Universitaire de Nîmes
Locations (2):
- France (2):
  - CHRU de Montpellier - Hôpital Lapeyronie, Montpellier
  - CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes